CLINICAL TRIAL: NCT02885233
Title: Evaluation of a Web-Based Fall Prevention Program on People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Michelle Cameron, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00015595
Record Dates: First submitted 2016-08-22; First posted 2016-08-31 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Multiple Sclerosis
Keywords: Fall Prevention; Multiple Sclerosis; Web-based education; Self-efficacy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free From Falls (Active Comparator): Subjects in the active group will participate in the Free From Falls Online Program consisting of 8 weekly 30 minute webinars providing education about risk factors for falls and fall prevention strategies; self-assessment exercises to evaluate understanding of the material; video-based exercise program targeting balance, posture, strength and flexibility to be performed at least 3 times per week; supplementary, downloadable printed material for both education and exercise; and a social forum to allow participants to interact with each other.
  Interventions: Behavioral: Free From Falls Online
- Waitlist (Placebo Comparator): Subjects in the waitlist control condition will receive an educational brochure developed by the National Multiple Sclerosis Society called "Minimizing Your Risk of Falls: A Guide for People with MS," which includes information on identifying risk factors for falling and fall risk management approaches with no exercise component; will inform their provider that they have fallen at least twice in the previous 2 months and discuss subsequent falls over the course of the 5-month study; and will be invited to participate in the Free From Falls Online Program at study completion.
  Interventions: Behavioral: Waitlist Control

INTERVENTIONS:
Behavioral: Free From Falls Online — Subjects in the active group will participate in the Free From Falls Online Program consisting of 8 weekly 30 minute webinars providing education about risk factors for falls and fall prevention strategies; self-assessment exercises to evaluate understanding of the material; video-based exercise program targeting balance, posture, strength and flexibility to be performed at least 3 times per week; supplementary, downloadable printed material for both education and exercise; and a social forum to allow participants to interact with each other.
  Arms: Free From Falls
Behavioral: Waitlist Control — Subjects in the waitlist control condition will receive an educational brochure developed by the National Multiple Sclerosis Society called "Minimizing Your Risk of Falls: A Guide for People with MS," which includes information on identifying risk factors for falling and fall risk management approaches with no exercise component; will inform their provider that they have fallen at least twice in the previous 2 months and discuss subsequent falls over the course of the 5-month study; and will be invited to participate in the Free From Falls Online Program at study completion.
  Arms: Waitlist

SUMMARY:
This study evaluates the effectiveness of a web-based fall prevention program called Free From Falls Online (FFFO) on people with multiple sclerosis.

DETAILED DESCRIPTION:
The overarching goal of this study is to evaluate the effectiveness and impact of an online self-management program for preventing falls among people with multiple sclerosis (PwMS). To accomplish this objective, the investigators have designed a web-based fall prevention program called Free From Falls Online (FFFO), based on the traditionally in-person program developed by the National Multiple Sclerosis Society. The specific aims of this study are three-fold: (1) to evaluate the effectiveness of an online fall prevention self-education program by comparing fall frequency between participants and controls; (2) evaluate the impact of FFFO by comparing patient reported measures of physical function, fatigue, self-efficacy, psychosocial illness impact, social participation and satisfaction, and perception of global health between participants and controls; (3) and to determine usability of and satisfaction with FFFO.

ELIGIBILITY:
Inclusion Criteria:

* MS of any type with no relapse in the previous month
* Self-reported history of 2 or more falls in the previous 2 months
* Ability to walk at least 100 meters with intermittent or unilateral constant assistance (Expanded Disability Severity Scale (EDSS) step <6.0)
* Daily access a computer and willingness to respond to a daily survey

Exclusion Criteria:

* Medical conditions that would preclude reliable participation or increases risk for injury during the program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
Difference in mean change in total falls between intervention and control arms | 5 months
  To determine if participation in FFFO is associated with decreased frequency of falls, subjects will be randomly assigned to either the active intervention group or the waitlist control group. All subjects will prospectively document the number and circumstances of their falls for 5 months through the use of an electronic survey, to include the 8 weeks of the active or control intervention and 3-month follow-up. The primary outcome will be the difference in fall frequency between active and control subjects.

SECONDARY OUTCOMES:
Difference in patient reported outcomes including physical function, fatigue, self efficacy, psychosocial illness impact, social participation and satisfaction, and perception of global health between intervention and control arms. | 5 months
  To determine if participation in FFFO is associated with improvement in patient reported outcomes, subjects will be randomly assigned to either the active intervention group or the waitlist control group. Outcomes will be measured through the use of the Patient Reported Outcomes Measurement Information System (PROMIS) which has been validated in people with multiple sclerosis. All subjects will complete the questionnaires at baseline, at 8 weeks and at 3 month follow-up. Scores will be compared between active and control subjects.
Quantitative assessment of the web-based program | 8 weeks
  To determine usability and satisfaction with FFFO, subjects in the active group will complete a computer-based questionnaire at the end of the program. The investigators will quantitatively evaluate participant assessment of the FFFO program through the use of a 5-point Likert scale.
Qualitative assessment of the web-based program | 8 weeks
  To determine usability and satisfaction with FFFO, subjects in the active group will complete a computer-based questionnaire at the end of the program. The investigators will qualitatively evaluate participant assessment of the FFFO program through the use of free-text responses.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle H Cameron, MD, Principal Investigator — Portland VA Medical Center
Locations (1):
- Oregon Health Sciences University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No